CLINICAL TRIAL: NCT00193882
Title: A Randomised Phase III Study in Advanced Oesophageal Cancer to Compare Quality of Life and Palliation of Dysphagia in Patients Treated With Radiotherapy vs ChemoRadiotherapy.
Brief Title: Advanced Oesophageal Cancer Study to Compare Quality of Life and Palliation of Dysphagia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 03.01; NCIC CTG ES.2 (Other: National Cancer Institute of Canada Clinical Trials Group); TGA 2004/83 (Other: Theraputic Goods of Australia); NHMRC 291103 (Other: National Health and Medical Research Council)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Esophagus Cancer
Keywords: Oesophageal; Dysphagia; Palliation; Quality of Life; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders | interventions — Cisplatin; Radiotherapy; Radiation; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Radiotherapy (Active Comparator): Radiotherapy alone
  Interventions: Radiation: Radiotherapy
- B: Chemo-radiotherapy (Experimental): Chemotherapy (Cisplatin + 5-Fluorouracil ) and Radiotherapy
  Interventions: Drug: Cisplatin; Radiation: Radiotherapy; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Cisplatin — 80mg/m2 IV day 1
  Other Names: Cisplatin Injection
  Arms: B: Chemo-radiotherapy
Radiation: Radiotherapy — 35 Gy in 15 fractions
  Other Names: Radiation; Radiation Therapy
Drug: 5-Fluorouracil — 800mg/m2/day IV days 1 - 4
  Other Names: DBL Flurouracil Injection BP, Efudix
  Arms: B: Chemo-radiotherapy

SUMMARY:
To compare the treatment of gullet cancer with radiotherapy alone and assess the advantage and toxicity of adding chemotherapy. The hypothesis to be tested is as follows: That the addition of chemotherapy to a short course of radiation treatment improves the proportion of patients who achieve relief of dysphagia and improves quality of life compared to radiation alone in patients with advanced oesophageal cancer.

DETAILED DESCRIPTION:
Prospective radical treatment trials in oesophageal cancer have shown responses in both radiotherapy alone and radiotherapy when combined with chemotherapy. Retrospective studies show a response in the palliative setting to relieve dysphagia. The response, durability and quality of life end points have not been previously fully documented. This will be addressed by this trial.

Dysphagia is the commonest presenting symptom due to local disease obstructing the oesophagus. Difficulty eating not only affects the patient's ability to maintain nutrition, but also impacts on all areas of quality of life. Relief of dysphagia becomes the highest priority for treatment.

At the time of developing this protocol there were no randomised trials comparing chemo-radiotherapy and radiotherapy in the palliative setting.

Few studies have prospectively assessed quality of life data for patients with oesophageal cancer, and although toxicity and survival data is available, there is no long-term data on quality of life. This trial will assess quality of life in a consecutive manner using a standardised self-reporting measure of quality of life, and compare quality of life across two groups having different treatments.

Eligible patients are those with proven carcinoma of the oesophagus who are deemed not suitable for definitive radical treatment due to the advanced nature of disease, presence of metastases or intercurrent illness, who have symptomatic dysphagia requiring loco-regional palliation.

Patients will be randomised to the following treatment options:

1. Radiotherapy Alone

   * 35 Gy in 15 fractions (Australia and New Zealand) or
   * 30 Gy in 10 fractions(Canada ONLY)
2. Chemo-Radiotherapy

   * 35 Gy in 15 fractions (Australia and New Zealand) or
   * 30 Gy in 10 fractions (Canada ONLY)
   * Cisplatin 80mg/m2 IV day 1 (or 20mg/m2/day IV days 1 - 4)
   * 5-Fluorouracil 800mg/m2/day IV days 1 - 4

Patients will have an initial baseline assessment then be followed up weekly during treatment, monthly for 1 year post treatment and then 3 monthly.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven Carcinoma of the oesophagus.
* Not a candidate for radical/curative treatment due to the advanced nature of the disease, presence of metastases, or intercurrent illness. (It should be noted that, patients with mediastinal nodes and no more distant disease maybe suitable for radical treatment).
* Symptomatic patients with dysphagia scores of ≥ 1 i.e. able to eat only some solids (see Mellow Scale appendix 1)
* Performance status ECOG ≤ 2
* Patients must begin treatment within 2 weeks of randomization.
* Patient is at least 18 years old.
* Adequate haematological function to undergo chemotherapy. Peripheral blood - Neutrophils > 1.5 x 10^9/L - Platelets > 100 x 10^9/L
* Adequate renal function, Creatinine - Calculated clearance ≥ 50 ml/min
* Patients capable of childbearing are using adequate contraception.
* Written informed consent of patient.

Exclusion Criteria:

* Previous mega-voltage external beam Radiotherapy or brachy-therapy delivered to the region of the chest.
* Synchronous active malignancies.
* Pregnant or lactating patients.
* Patients unfit for any treatment component.
* Tracheo-oesophageal fistula.
* Stents in situ.
* Previous chemotherapy for Oesophageal Cancer
* CT scan of thorax and abdomen more than 8 weeks prior to randomization
* Full Blood Count, Biochemistry (including creatinine) and creatinine clearance more than 2 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2003-07-07; Primary Completion 2012-03-21 (Actual); Study Completion 2013-06-18 (Actual)

PRIMARY OUTCOMES:
Relief of dysphagia | This will be measured at nine weeks after the start of radiotherapy and must be maintained at the next review 4 weeks thereafter.

SECONDARY OUTCOMES:
Dysphagia progression free survival. | This will be measured from randomisation to the time of first progression of dysphagia.
Quality of Life differences post treatment and at 3 months and 6 months. | post treatment and at 3 months and 6 months.
Acute and late toxicity. | Interim analyses planned at 110 pateints. Final analyses will occur after 5 years.
Survival. | Interim analyses planned at 110 pateints. Final analyses will occur after 5 years.
Time to achieving any response in dysphagia after treatment as measured by an improvement of at least 1 point on the 5 point dysphagia scale. | Interim analyses planned at 110 pateints. Final analyses will occur after 5 years.
Number of patients receiving secondary treatment (radiation, chemotherapy or stenting). | Interim analyses planned at 110 pateints. Final analyses will occur after 5 years.
Time to achieving a complete response i.e. dysphagia score of 0. | Interim analyses planned at 110 pateints. Final analyses will occur after 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Penniment, FRANZCR, Study Chair — Royal Adelaide Hopsital
Locations (25):
- Australia (15):
  - Liverpool Hospital, Liverpool, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Premion - Wesley, Auchenflower, Queensland
  - Royal Brisbane Hospital, Herston, Queensland
  - Radiation Oncology - Mater Centre, South Brisbane, Queensland
  - North Queensland Oncology Service, Townsville, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Peter MacCallum - Box Hill Hospital, Box Hill, Victoria
  - Peter MacCallum - Moorrabbin, East Bentleigh, Victoria
  - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Canada (8):
  - Cross Cancer Centre, Edmonton, Alberta
  - Cancer Care Manitoba Winnipeg, Winnipeg, Manitoba
  - Saint John Regional Hospital - Atlantic Health Sci, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cancer Centre of Southeastern Ontario Kingston, Kingston, Ontario
  - Grand River Cancer Centre, Kitchener, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hotel-Dieu de Quebec, Québec
- Christchurch Hospital, Christchurch, New Zealand
- Princess Royal Hospital, Hull, United Kingdom

REFERENCES:
- [Derived] Penniment MG, De Ieso PB, Harvey JA, Stephens S, Au HJ, O'Callaghan CJ, Kneebone A, Ngan SY, Ward IG, Roy R, Smith JG, Nijjar T, Biagi JJ, Mulroy LA, Wong R; TROG 03.01/CCTG ES.2 group. Palliative chemoradiotherapy versus radiotherapy alone for dysphagia in advanced oesophageal cancer: a multicentre randomised controlled trial (TROG 03.01). Lancet Gastroenterol Hepatol. 2018 Feb;3(2):114-124. doi: 10.1016/S2468-1253(17)30363-1. Epub 2017 Dec 14. PMID 29248399
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au